CLINICAL TRIAL: NCT05460689
Title: A Randomized Controlled Trial to Evaluate the Effectiveness of a mHealth Application as a Family Educational and Supportive Tool in Children Tonsillectomy and/or Adenoidectomy Perioperative Process Compared to Standard Care
Brief Title: Effectiveness of a mHealth Application as a Family Supportive Tool in Pediatric Otolaryngology Perioperative Process
Acronym: TONAPP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 03/2022
Record Dates: First submitted 2022-07-11; First posted 2022-07-15 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: TONSILLECTOMY
Keywords: MHealth; Tonsillectomy; Education
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartphone Application (Experimental): mHealth App provided to caregivers of children undergoing tonsillectomy and/or adenoidectomy
  Interventions: Other: M-HEALTH APP
- standard support (Sham Comparator): Information provided by nurses and physician orally or through printed booklets.
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: M-HEALTH APP — The intervention group will have in use a mHealth App for education and support of caregivers of children undergoing tonsillectomy and/or adenoidectomy in the perioperative process. An out-patient nurse will be in charge of instructing intervention group participants to mHealth App use and content options. The mHealth App will be available for intervention group families from the day of pre-admission visits to the 7th day post surgery or follow up visit.
  Arms: Smartphone Application
Other: Standard Care — The control group will receive information and education provided by nurses and physician in the preoperative visits and during hospitalization. Information and education will be provided orally or through printed booklets.
  Arms: standard support

SUMMARY:
Tonsillectomy and/or adenoidectomy are common surgeries in children. Authors report how distressed children and their families are by perioperative processes. Fear of the unknown can put a strain on the preoperative period, while pain and other possible complications such as fever, vomiting, restricted oral feeding or bleeding can create difficulties in postoperative home management. Parental anxiety has been found to worsen the perception of pain, perioperative discomfort and recovery of operated children. Providing children and families with preparation for hospitalisation, surgery and postoperative home management has been shown to improve perioperative outcomes. However, not all individuals can understand and benefit from the information provided by healthcare professionals: higher levels of anxiety in the perioperative process have been associated with individuals with low health literacy. Furthermore, unmet information needs may lead parents to expose themselves to health-related misinformation through autonomous investigations on the Web and common social media resources. Patient- and family-centred education and support is a complex and time-consuming care practice, while some surgeries such as tonsillectomy are characterised by short hospitalisations that limit the amount of time health professionals can devote to this programme. Health systems have been testing different types of formats, content and ways of delivering health information/education in order to meet the requirements of clients, time availability and effectiveness. MHealth apps in particular are an essential element of e-health and consist of medical information that is available via mobile phones or other wireless devices and can be used by patients or health professionals. Their use is growing and evolving into a variety of functionalities and positive outcomes related to improving the wellbeing of individuals, including diagnostics and clinical decision-making; interventions on healthy behaviours and lifestyles; patient disease management and self-care. Findings from literature highlight the need for further randomised controlled trials to confirm positive results.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers of children aged 2-10 scheduled for tonsillectomy and/or adenoidectomy with or without tympanostomy tubes insertion;
* Caregivers who are capable of oral and written communication without any impairment;
* Caregivers who guarantee access to a smartphone and internet connection.

Exclusion Criteria:

* Caregivers with cognitive deficits;
* Caregivers of children with cognitive impairment
* Caregivers with visual impairment;
* Caregivers of children affected by chronic pain;
* Caregivers of children who had another surgery operation in the previous month.
* Caregivers who never used at least one smart phone application

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2022-12-16 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Between groups difference in preoperative primary child caregiver state anxiety (T2) | 5 minutes before heading to the operating theatre
  Differences between intervention and control groups in preoperative primary child caregiver state anxiety, measured through the State-Trait Anxiety Inventory form Y questionnaire (T2). The questionnaire consists of two self-report scales for measuring state anxiety and trait anxiety. The S-Anxiety scale (STAI Form Y-1) consists of twenty statements that evaluate how the respondent feels "now, at this moment," on a 4 items Likert scale, from "not at all" to "very much"; the T-Anxiety scale (STAI Form Y-2) consists of twenty statements that evaluate how the respondent feels "generally" on a 4-point Likert scale from "almost never" to "almost always". Total scores range from 20 to 80 points with lower scores indicate higher trait and state anxiety.

SECONDARY OUTCOMES:
Between groups difference in state anxiety assessment at post-operative follow up (T3) | 7 days after surgery
  Differences between intervention and control groups in post-operative primary child caregiver state anxiety, measured through the State-Trait Anxiety Inventory form Y questionnaire (T3). The questionnaire consists of two self-report scales for measuring state anxiety and trait anxiety. The S-Anxiety scale (STAI Form Y-1) consists of twenty statements that evaluate how the respondent feels "now, at this moment," on a 4 items Likert scale, from "not at all" to "very much"; the T-Anxiety scale (STAI Form Y-2) consists of twenty statements that evaluate how the respondent feels "generally" on a 4-point Likert scale from "almost never" to "almost always". Total scores range from 20 to 80 points with lower scores indicate higher trait and state anxiety.caregiver state anxiety will be measured through the State-Trait Anxiety Inventory form Y questionnaire in the surgical department, before heading to the operating theatre on the day of surgery (T1).
Between groups difference in state anxiety from enrollment and preoperative evaluations (T0 vs T2) | 5 minutes after enrolment / 5 minutes before heading to the operating theatre
  Differences between intervention and control groups primary child caregiver state anxiety from enrollment and preoperative evaluations, measured through the State-Trait Anxiety Inventory form Y questionnaire. The questionnaire consists of two self-report
Between groups difference in state anxiety from enrollment and post-operative follow up evaluations (T0 vs T3) | 5 minutes after enrolment / 7 days after surgery
  Differences between intervention and control groups primary child caregiver state anxiety from enrollment and post-operative follow up evaluations, measured through the State-Trait Anxiety Inventory form Y questionnaire. The questionnaire consists of two self-report scales for measuring state anxiety and trait anxiety. The S-Anxiety scale (STAI Form Y-1) consists of twenty statements that evaluate how the respondent feels "now, at this moment," on a 4 items Likert scale, from "not at all" to "very much"; the T-Anxiety scale (STAI Form Y-2) consists of twenty statements that evaluate how the respondent feels "generally" on a 4-point Likert scale from "almost never" to "almost always". Total scores range from 20 to 80 points with lower scores indicate higher trait and state anxiety.
Between groups difference in preoperative children distress (T2) | 5 minutes before heading to the operating theatre
  Difference between the intervention and control group in children distress assessed by surgery nurses in the surgical ward through the modified Yale Preoperative Anxiety Scale (mYPAS). The mYPAS consists of 27 items exploring five domains such as activity, emotional expressivity, state of arousal, vocalisation and use of caregivers. Scores range from 23.33 to 100, with higher scores indicating higher levels of anxiety.
Between groups difference in parents' preparation for hospitalization and surgery (T1) | Within 30 minutes after the admission in the surgery ward
  The difference between the intervention and control group in parents' preparation for hospitalization and surgery evaluated by nurses through documents missing at hospital admission for surgery (number of documents missing) and surgery preparation items missing such as total body hygiene; nail polish removal and fasting (number of preparations items missing)
Between groups difference in the social and health impact of the introduction of an mHealth App | 7 days after surgery
  The differences between the intervention and control group in the social and health impact of the introduction of an mHealth App, measured through an ad hoc questionnaire on the day of follow up visit

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Cassone, RN, BSN MES, Study Chair — Institute for Maternal and Child Health IRCCS Burlo Garofolo; Raffaella Dobrina, RN, BSN MES, Principal Investigator — Institute for Maternal and Child Health IRCCS Burlo Garofolo
Locations (1):
- Institute for Maternal and Child Health - IRCCS "Burlo Garofolo", Trieste, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dobrina R, Cassone A, Dal Cin M, Ronfani L, Giangreco M, Schreiber S, Zanchiello S, Starec A, Brunelli L, Brumatti LV, Bicego L. Study protocol for a randomised controlled trial to determine the effectiveness of a mHealth application as a family supportive tool in paediatric otolaryngology perioperative process (TONAPP). Trials. 2023 May 25;24(1):355. doi: 10.1186/s13063-023-07376-z. PMID 37231477